CLINICAL TRIAL: NCT01016249
Title: Nebulized 5% Hypertonic Saline for Infirmary Treatment of Acute Infant Bronchiolitis: A Randomized Trial
Brief Title: Nebulized 5% Hypertonic Saline for the Treatment of Bronchiolitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Dr Khalid Al Ansari, Hamad Medical Corporation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: #7055
Record Dates: First submitted 2009-11-18; First posted 2009-11-19 (Estimated); Last update posted 2009-11-19 (Estimated); Status verified 2009-11

CONDITIONS: Bronchiolitis
Keywords: Bronchiolitis, Viral; An acute inflammation of the upper RESPIRATORY TRACT
MeSH Terms: conditions — Bronchiolitis; Bronchiolitis, Viral | interventions — Saline Solution, Hypertonic; Epinephrine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment 1. 5% Saline + Epinephrine (Active Comparator): Nebulization with 4ml of 5% saline mixed with 1.5 ml of epinephrine every 4 hours thereafter until ready for discharge. Immediately before nebulization, just after, and 2 hours after, the following measurements were collected for each patients: bronchiolitis severity score, oxygen saturation on room air, and heart rate.
  Interventions: Drug: Treatment 1. (5% Hypertonic saline + Epinephrine)
- Treatment 3. 3% Saline + Epinephrine (Other): Nebulization with 4ml of 3% saline mixed with 1.5 ml of epinephrine every 4 hours thereafter until ready for discharge. Immediately before nebulization, just after, and 2 hours after, the following measurements were collected for each patients: bronchiolitis severity score, oxygen saturation on room air, and heart rate.
  Interventions: Drug: Treatment 3. (3% Hypertonic saline + Epinephrine)
- Treatment 2 . 0.9% Saline + Epinephrine (Other): Nebulization with 4ml of 0.9% saline mixed with 1.5 ml of epinephrine every 4 hours thereafter until ready for discharge. Immediately before nebulization, just after, and 2 hours after, the following measurements were collected for each patients: bronchiolitis severity score, oxygen saturation on room air, and heart rate.
  Interventions: Drug: Treatment 2. (Normal saline + Epinephrine)

INTERVENTIONS:
Drug: Treatment 1. (5% Hypertonic saline + Epinephrine) — Nebulization of 4ml 5% saline mixed with 1.5 ml of epinephrine on enrollment and every 4 hours thereafter until ready for discharge.
  Other Names: 5% Hypertonic saline
  Arms: Treatment 1. 5% Saline + Epinephrine
Drug: Treatment 3. (3% Hypertonic saline + Epinephrine) — Nebulization of 4ml 3% saline mixed with 1.5 ml of epinephrine on enrollment and every 4 hours thereafter until ready for discharge.
  Other Names: 3% Hypertonic saline
  Arms: Treatment 3. 3% Saline + Epinephrine
Drug: Treatment 2. (Normal saline + Epinephrine) — Nebulization of 4ml 0.9% saline mixed with 1.5 ml of epinephrine on enrollment and every 4 hours thereafter until ready for discharge.
  Other Names: Normal saline
  Arms: Treatment 2 . 0.9% Saline + Epinephrine

SUMMARY:
The investigators reasoned that a hypertonic saline concentration higher than 3% could be safe and more efficacious in the treatment of bronchiolitis, alleviating severe symptoms and preventing the need for hospitalization in some instances.

DETAILED DESCRIPTION:
We conducted a double blind, randomized, parallel-group clinical trial to compare the efficacy and safety of hypertonic saline 3% and 5% versus normal saline for the treatment of acute bronchiolitis.

The study was conducted in the short stay unit of the Pediatric Emergency Center of Hamad General Hospital, the only pediatric emergency facility in the State of Qatar. The Center serves an average of 200,000 patients annually and manages 42 beds in the short stay unit. Patients admitted to the unit were assessed at least every 6 hours by a pediatrician to determine readiness for discharge. The length of stay in the unit for bronchiolitis range from 6 to 168 hours.

Infants aged ≤18 months presenting to the unit for the treatment of moderate-severe viral bronchiolitis were eligible for the study. Moderate-severe bronchiolitis required having a prodromal history consistent with viral upper respiratory tract infection followed by wheezing and/or crackles on auscultation and a Wang bronchiolitis severity score of ≥ 4 on presentation.

Patients were excluded from the study if they had one or more of the following characteristics: Born preterm ≤34 weeks gestation, previous history of wheezing, steroid use within 48 hours of presentation, obtundation and progressive respiratory failure requiring ICU admission, history of apnea with in 24 hours before presentation, oxygen saturation ≤ 85% on room air at the time of recruitment, history of a diagnosis of chronic lung disease, congenital heart disease, or immunodeficiency.

The six attending physicians who covered the 18 beds in the respiratory section of the short stay unit were trained in scoring and its practical application on our bronchiolitis patients in the unit before the study began.

Written and informed consent, was sought from one of the parents or legal guardians for eligible patients as soon as the patient was admitted to the unit. The study was approved by the hospital institutional review board.

Patients were examined on presentation and those requiring further treatment or observation were admitted to the short stay unit. Those with bronchiolitis were assessed for study eligibility within 2 hours of the initial physician assessment. Patients for whom consent was obtained underwent plain chest radiography and nasopharyngeal swabs were taken for RSV detection (RSV Respi-Strip, Coris Bioconcept, Gembloux, Belgium). Then a computer-generated list of random numbers was used by the enrolling physicians in consecutive order to identify a sealed envelope containing one of three codes identifying one of three different bags of 500 mL of sterilely-prepared blinded study solution, made fresh each morning by a pharmacist blinded to patient assignment.Patients received the study nebulization mixed with 1.5 ml of epinephrine in a double blinded fashion on enrollment and every 4 hours thereafter until they were ready for discharge.Additional nebulized epinephrine 5ml delivered the same way was administered with blinded study solution at a maximum frequency of every hour and additional treatment (e.g., supplementary oxygen, hydration) given at the discretion of the treating physician. Patients were withdrawn from the study if oxygen saturation within 30 min after nebulization fell below 85% on room air or clinical deterioration was determined to warrant transfer to the pediatric intensive care unit. Patients were discharged when the treating physician determined the patient did not need supplementary oxygen, was feeding adequately without intravenous fluids, and had minimal or absent wheezing, crackles, and chest retractions provided he/she had an oxygen saturation ≥ 94% and severity score < 4 on discharge.

At discharge, patients were sent home with albuterol metered-dose inhalers . Follow-up by study nurse by telephone was mandatory daily, for one week after discharge. The patient could return to the pediatric emergency center earlier if desired or needed.

ELIGIBILITY:
Inclusion Criteria:

* Infants aged ≤ 18 months presenting to the unit for the treatment of moderate-severe viral bronchiolitis were eligible for the study.
* Moderate-severe bronchiolitis required having a prodromal history consistent with viral upper respiratory tract infection followed by wheezing and/or crackles on auscultation and a Wang bronchiolitis severity score of ≥ 4 on presentation.

Exclusion Criteria:

Patients were excluded from the study if they had one or more of the following characteristics:

* Born preterm ≤ 34 weeks gestation,
* Previous history of wheezing,
* Steroid use within 48 hours of presentation,
* Obtundation and progressive respiratory failure requiring ICU admission,
* History of apnea with in 24 hours before presentation,
* Oxygen saturation ≤ 85% on room air at the time of recruitment,
* History of a diagnosis of chronic lung disease,
* Congenital heart disease, or
* Immunodeficiency.

Ages: 1 Day to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 187 (Actual)
Dates: Start 2007-04; Primary Completion 2008-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Mean pre-nebulization bronchiolitis severity score for each treatment group at 48 hours | 2 years

SECONDARY OUTCOMES:
The treatments' severity scores at 24 hours and trend over time to 72 hours, 2 hours-post-nebulization severity scores trending over time, as well as safety measures | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Khalid M. Al-Ansari, FRCPC,FAAP, Principal Investigator — Hamad Medical Corporation, Weill Cornell Medical College
Locations (1):
- Pediatric Emergency Center, Al-Saad, Doha, Baladīyat ad Dawḩah, Qatar

REFERENCES:
- [Derived] Al-Ansari K, Sakran M, Davidson BL, El Sayyed R, Mahjoub H, Ibrahim K. Nebulized 5% or 3% hypertonic or 0.9% saline for treating acute bronchiolitis in infants. J Pediatr. 2010 Oct;157(4):630-4, 634.e1. doi: 10.1016/j.jpeds.2010.04.074. Epub 2010 Jun 19. PMID 20646715